CLINICAL TRIAL: NCT02720848
Title: A Randomized Clinical Trial of a Novel Stiffening Wire to Increase Depth of Insertion During Double and Single Balloon Enteroscopy
Brief Title: Double/Single Balloon Enteroscopy Stiffening Wire RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 107609
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Small Intestine Problem
Keywords: double-balloon enteroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stiffening wire (Experimental): A stiffening wire inserted into the instrument channel of the double/single balloon enteroscope will be used.
  Interventions: Device: Stiffening wire
- Standard technique (Active Comparator): The double/single balloon enteroscope will be used without the stiffening wire as per standard technique.
  Interventions: Device: Standard technique

INTERVENTIONS:
Device: Stiffening wire — The stiffening wire will be inserted into the double/single balloon enteroscope.
  Arms: Stiffening wire
Device: Standard technique — The double/single balloon enteroscope will be used without the stiffening wire as per standard technique.
  Arms: Standard technique

SUMMARY:
This is a randomized clinical trial examining the use of a stiffening wire to increase depth of maximal insertion during double and single balloon enteroscopy.

DETAILED DESCRIPTION:
BACKGROUND Small bowel endoscopy has undergone a paradigm shift in the past decade. Prior to this, the small bowel was considered a 'black hole' due to our inability to visualize it endoscopically and the limited sensitivity of radiologic studies. This all changed with the development of capsule endoscopy, which gave physicians the ability to visualize the full length of the small bowel. Although widely considered a great leap forward, video capsule endoscopy is limited by its inability to perform any form of endoscopic intervention. Thus, something was needed to biopsy and treat the abnormalities detected with capsule endoscopy. Double balloon enteroscopy (DBE) was invented in Japan in 2001. Using an overtube and two inflatable balloons, DBE enabled deep intubation of the small bowel through a series of push and pull maneuvers to accordion the small bowel over the overtube. This procedure proved highly successful in the diagnosis and treatment of small bowel diseases. Subsequently, single balloon enteroscopy (SBE) was developed consisting of a single overtube balloon. Collectively, these techniques are called balloon assisted enteroscopy.

Balloon assisted enteroscopy can be performed using an antegrade (through the mouth) or retrograde (through the anus) approach. The two approaches are considered complimentary since the antegrade approach enables visualization of the proximal and mid small bowel while the distal portion is seen with the retrograde approach. Complete enteroscopy, or visualization of the entire small intestine, occurs when an antegrade enteroscopy is performed and the tattoo left at the depth of maximal insertion is reached during a subsequent retrograde procedure. Although considered to be the gold standard for enteroscopy, this is rarely achieved outside of expert centres in Japan. The reason for this is because of loop formation in the small intestine, commonly referred to as looping (Figure 1). Looping typically worsens as the depth of insertion increases and eventually prevents forward migration of the enteroscope.

Looping is not unique to enteroscopy and is a common problem encountered during colonoscopy. During colonoscopy, loops can be removed, by pulling back and torqueing the colonoscope. However, the loop often reforms when the colonoscope is pushed forward again. To counter this problem, colonoscopes have been developed with adjustable stiffness that can be changed during the procedure (Olympus Inc., Tokyo, Japan). Using this feature, the loop can be removed and the colonoscope stiffened prior to pushing forward to prevent loop reformation.

Although variable stiffness is available in colonoscopes, the same technology cannot be incorporated into enteroscopes due to its much thinner diameter. Recently, an enteroscopy stiffening wire has been developed by Zutron Medical LLC (Kansas, USA). This through the scope wire can be inserted as needed to increase the stiffness of the enteroscope. In theory, this should improve the performance of DBE/SBE and translate into deeper insertion although this has never been investigated. The objective of this randomized clinical trial is to answer this question.

STUDY DESIGN

This is a single centre randomized clinical trial assessing whether a stiffening wire increases the depth of maximal insertion during DBE/SBE. Due to the nature of the procedure, blinding of the endoscopist is impossible. This is because even if a placebo wire is used, the enteroscope feels sufficiently different to enable unmasking. To mitigate the risk of bias, the enteroscopy will be recorded and outcomes assessed in a blinded fashion using the recorded video. Randomization will be in blocks of varying sizes and performed using sequentially labelled sealed envelopes.

STUDY INTERVENTION

1. After fasting overnight, sedation is given at the start of the procedure. This consists of either Propofol administered by an anesthetist or midazolam and fentanyl administered by the endoscopist.
2. The enteroscope is inserted into the mouth, down the esophagus, though the stomach, and into the duodenum.
3. Once in the small bowel, a series of push and pull maneuvers are used as previously described (1). Each set of maneuvers is called a cycle.
4. Cycles are repeated until looping prevents any further forward movement and the depth of maximal insertion is reached. In the study, depth of maximal insertion 1 will be defined as a lack of forward movement after 3 consecutive cycles.
5. When the depth of maximal insertion 1 has been reached, a small mark will be made on the wall of the small bowel by sucking mucosa into the enteroscope (ie. suction mark) or using biopsy forceps to create a 3 mm disruption in the mucosa. A virtual mark will also be made on the endoscopy video.
6. Those randomized to the stiffening wire will insert the wire and attempt to proceed deeper. The technique for each cycle is the same as in step 3 and does not change with the presence of the wire.
7. Those randomized to no stiffening wire will attempt to proceed deeper using standard technique.
8. The procedure will continue until there is no forward movement after 3 consecutive cycles. If the enteroscope was able to proceed past depth of maximal insertion 1, a suction/biopsy forceps mark will be made and a virtual mark recorded on the endoscopy video to denote depth of maximal insertion 2. If the enteroscope was not able to proceed past depth of maximal insertion 1, no further marks will be made.
9. On withdrawal of the enteroscope, care will be taken by the endoscopist to ensure any suction/biopsy forceps marks are clearly visible on the video.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing antegrade DBE/SBE.

Exclusion Criteria:

* Age < 18
* Prior surgery involving resection of the esophagus, stomach, or small bowel
* Suspected stricture or mass in any part of the gastrointestinal tract
* Failure to obtain informed consent from the patient or substitute decision maker
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Distance gained beyond depth of maximal insertion 1 | Measured once at the time of endoscopy
  Defined as the distance between depth of maximal insertion 1 and depth of maximal insertion 2. In cases where there is no depth of maximal insertion 2, a value of zero will be assigned. Distance will be measured using the fold counting method as follows: distance = # fold x 0.904 cm/fold.

SECONDARY OUTCOMES:
Final depth of insertion | Measured once at the time of endoscopy
  Defined as the distance between depth of maximal insertion 2 (or depth of maximal insertion 1 if primary outcome = 0) and the pylorus. Distance will be measured using the fold counting method.
Small bowel diagnostic rate | Measured once at the time of endoscopy
  Small bowel diagnosis (dichotomous variable, yes/no) is defined as the visualization of a small bowel abnormality, such as an angioectasia, Crohn's disease, stricture, polyp, mass, or foreign body). Red spots are not included.
Small bowel intervention rate | Measured once at the time of endoscopy
  Small bowel therapeutics (dichotomous variable, yes/no) is defined as the application of endoscopic intervention to a small bowel abnormality, such as biopsy of a polyp/mass/ulcer, APC, dilation, polypectomy, or foreign body retrieval.
Patient comfort survey | Measured once at the time of endoscopy
  a. To be completed after the procedure in the recovery room using a visual analogue scale (1=no pain, 10=severe pain). Patients will be assessed for intraprocedural and postprocedural pain.
Serious Adverse events | Measured once at the time of endoscopy
  Perforation, bleeding requiring blood transfusion or hospital admission, pancreatitis, aspiration, significant hypotension (systolic blood pressure < 80 mmHg), hypoxia (oxygen saturation < 85%), or bradycardia (heart rate < 45 beats per minute). Assessed on day 0 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sey, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Yamamoto H, Sekine Y, Sato Y, Higashizawa T, Miyata T, Iino S, Ido K, Sugano K. Total enteroscopy with a nonsurgical steerable double-balloon method. Gastrointest Endosc. 2001 Feb;53(2):216-20. doi: 10.1067/mge.2001.112181. PMID 11174299
- [Background] Yamamoto H, Kita H, Sunada K, Hayashi Y, Sato H, Yano T, Iwamoto M, Sekine Y, Miyata T, Kuno A, Ajibe H, Ido K, Sugano K. Clinical outcomes of double-balloon endoscopy for the diagnosis and treatment of small-intestinal diseases. Clin Gastroenterol Hepatol. 2004 Nov;2(11):1010-6. doi: 10.1016/s1542-3565(04)00453-7. PMID 15551254
- [Background] May A, Nachbar L, Ell C. Double-balloon enteroscopy (push-and-pull enteroscopy) of the small bowel: feasibility and diagnostic and therapeutic yield in patients with suspected small bowel disease. Gastrointest Endosc. 2005 Jul;62(1):62-70. doi: 10.1016/s0016-5107(05)01586-5. PMID 15990821
- [Background] Hartmann D, Eickhoff A, Tamm R, Riemann JF. Balloon-assisted enteroscopy using a single-balloon technique. Endoscopy. 2007 Feb;39 Suppl 1:E276. doi: 10.1055/s-2007-966616. Epub 2007 Oct 24. No abstract available. PMID 17957636
- [Background] Kawamura T, Yasuda K, Tanaka K, Uno K, Ueda M, Sanada K, Nakajima M. Clinical evaluation of a newly developed single-balloon enteroscope. Gastrointest Endosc. 2008 Dec;68(6):1112-6. doi: 10.1016/j.gie.2008.03.1063. Epub 2008 Jul 2. PMID 18599052
- [Background] Domagk D, Mensink P, Aktas H, Lenz P, Meister T, Luegering A, Ullerich H, Aabakken L, Heinecke A, Domschke W, Kuipers E, Bretthauer M. Single- vs. double-balloon enteroscopy in small-bowel diagnostics: a randomized multicenter trial. Endoscopy. 2011 Jun;43(6):472-6. doi: 10.1055/s-0030-1256247. Epub 2011 Mar 7. PMID 21384320
- [Background] Efthymiou M, Desmond PV, Brown G, La Nauze R, Kaffes A, Chua TJ, Taylor AC. SINGLE-01: a randomized, controlled trial comparing the efficacy and depth of insertion of single- and double-balloon enteroscopy by using a novel method to determine insertion depth. Gastrointest Endosc. 2012 Nov;76(5):972-80. doi: 10.1016/j.gie.2012.06.033. Epub 2012 Sep 12. PMID 22980289
- [Background] May A, Farber M, Aschmoneit I, Pohl J, Manner H, Lotterer E, Moschler O, Kunz J, Gossner L, Monkemuller K, Ell C. Prospective multicenter trial comparing push-and-pull enteroscopy with the single- and double-balloon techniques in patients with small-bowel disorders. Am J Gastroenterol. 2010 Mar;105(3):575-81. doi: 10.1038/ajg.2009.712. Epub 2010 Jan 5. PMID 20051942
- [Background] Takano N, Yamada A, Watabe H, Togo G, Yamaji Y, Yoshida H, Kawabe T, Omata M, Koike K. Single-balloon versus double-balloon endoscopy for achieving total enteroscopy: a randomized, controlled trial. Gastrointest Endosc. 2011 Apr;73(4):734-9. doi: 10.1016/j.gie.2010.10.047. Epub 2011 Jan 26. PMID 21272875
- [Background] Yamamoto H, Kita H. Enteroscopy. J Gastroenterol. 2005 Jun;40(6):555-62. doi: 10.1007/s00535-005-1645-5. PMID 16007388
- [Derived] Archer M, Liu E, McDonald C, Yan B, Jairath V, Sey M. A randomized controlled trial of a through-the-scope stiffening wire to increase the depth of insertion during double-balloon enteroscopy. Gastrointest Endosc. 2025 Jun;101(6):1197-1200. doi: 10.1016/j.gie.2024.11.037. Epub 2024 Nov 26. PMID 39608590